CLINICAL TRIAL: NCT00322621
Title: Maintenance of Effect of Duloxetine 60 mg Once Daily in Patients With Diabetic Peripheral Neuropathic Pain
Brief Title: Maintenance of Effect of Duloxetine in Patients With Diabetic Peripheral Neuropathic Pain (DPNP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10258; F1J-MC-HMEM (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2009-12-18 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride

ARMS (1):
- Duloxetine (Experimental): All subjects receive 30 mg once daily (QD), by mouth (per os - PO) for 1 week followed by duloxetine 60 mg QD, PO for 7 weeks, then maintenance at 60 mg QD, PO for responders to 6 months and rescue at 120 mg QD, PO for non-responders to 6 months. Patients beginning maintenance at the 60 mg QD dose could be increased to the 120 mg QD level if they did not maintain appropriate level of response throughout the maintenance period.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine
  Other Names: LY248686; Cymbalta

SUMMARY:
To determine if duloxetine 60 mg once daily can work up to 6 months in treating pain from Diabetic Neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Have pain due to bilateral peripheral neuropathy caused by Type I or Type II diabetes with the pain beginning in the feet and present for at least 6 months.
* May not be pregnant and agree to utilize medically acceptable and reliable means of birth control during participation in the study.
* Score of 4 or greater on the Brief Pain Inventory on the 24-hour average pain item.

Exclusion Criteria:

* History of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Serious or unstable cardiovascular, hepatic (acute liver injury such as hepatitis or severe cirrhosis),kidney, respiratory, or blood disorder, seizure disorder, problems with peripheral vascular disease, or other medical conditions or psychiatric conditions that would hinder your participation or be likely to lead to hospitalization during the course of the study.
* Taking monoamine oxidase inhibitor (MAOI) within 14 days of starting the study or the potential need to take during or within 5 days after discontinuation from the study.
* Treatment with fluoxetine within 30 days of starting the study.
* Unstable blood sugar control and uncontrolled or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (19):
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fortaleza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto Alegre
- France (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Annecy
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dijon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Narbonne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nevers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chemitz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Münster
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Schkeuditz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Würzburg
- Italy (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Perugia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome

REFERENCES:
- [Result] Skljarevski V, Desaiah D, Zhang Q, Chappell AS, Detke MJ, Gross JL, Ziegler D. Evaluating the maintenance of effect of duloxetine in patients with diabetic peripheral neuropathic pain. Diabetes Metab Res Rev. 2009 Oct;25(7):623-31. doi: 10.1002/dmrr.1000. PMID 19637208
- [Derived] Hall JA, Wang F, Oakes TM, Utterback BG, Crucitti A, Acharya N. Safety and tolerability of duloxetine in the acute management of diabetic peripheral neuropathic pain: analysis of pooled data from three placebo-controlled clinical trials. Expert Opin Drug Saf. 2010 Jul;9(4):525-37. doi: 10.1517/14740338.2010.484418. PMID 20465525
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was a 5-9 day Screening Phase. Study Period II was an 8 week Acute Therapy Phase. Study Period III was a 26 week Maintenance and Rescue Therapy Phase. Study Period IV was a 2 week Taper Phase.
Groups:
- Acute Phase: All subjects receive 30 milligrams (mg) duloxetine once daily (QD), by mouth (PO) for 1 week followed by duloxetine 60 mg QD, PO for 7 weeks, then maintenance at 60 mg QD, PO for responders to 6 months and rescue at 120 mg QD, PO for non-responders to 6 months.
- Maintenance Arm: Duloxetine: 60 milligrams once daily.
- Rescue Arm: Duloxetine: 120 milligrams once daily.
Period: Period II - Acute Therapy Phase
Arm/Group | Acute Phase | Maintenance Arm | Rescue Arm
Started | 216 | 0 | 0
Completed | 184 | 0 | 0
Not Completed | 32 | 0 | 0
Not completed — Adverse Event | 20 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Period III - Maintenance / Rescue Phase
Arm/Group | Acute Phase | Maintenance Arm | Rescue Arm
Started | 0 | 115 | 69
Completed | 0 | 86 | 33
Not Completed | 0 | 29 | 36
Not completed — Adverse Event | 0 | 14 | 5
Not completed — Lack of Efficacy | 0 | 4 | 24
Not completed — Withdrawal by Subject | 0 | 7 | 1
Not completed — Protocol Violation | 0 | 2 | 5
Not completed — Death | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acute Phase
Number analyzed (Participants) | 216
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 112
Region of Enrollment [Number; unit: participants]
  France | 43
  Brazil | 66
  Germany | 66
  Italy | 41
Duration of Diabetes [Number; unit: participants]
  <=2 years | 78
  >2 years | 138
Duration of Neuropathic Pain [Number; unit: participants]
  <=1 year | 38
  >1 year | 178
Race/Ethnicity [Number; unit: participants]
  Caucasian | 173
  West Asian | 33
  African | 6
  Hispanic | 4
Type of Diabetes Mellitus [Number; unit: participants]
  Type 1 | 12
  Type 2 | 204
Brief Pain Inventory 24-Hour Average Pain Severity [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.88 (1.45)
Height at Visit 1 (Week -1) [Mean (Standard Deviation); unit: centimeters (cm)] | 166.7 (10.39)
Weight at Visit 2 (Week 0) [Mean (Standard Deviation); unit: kilograms (kg)] | 84.0 (18.36)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 8) in Brief Pain Inventory (BPI) 24-hour Average Pain Item Score at Week 34 Endpoint
Description: Maintenance effect of duloxetine 60 mg in patients with diabetic peripheral neuropathic pain (DPNP) was assessed by the change in BPI 24-hour average pain item score from baseline of the maintenance therapy arm (week 8) to 34 week endpoint in patients who achieved at least a 30 percent reduction on the BPI 24-hour average pain item after 8 weeks of acute therapy (Acute Therapy Phase). BPI is a self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 8), Week 34
Population: Patients entering maintenance phase on duloxetine 60 mg QD. Endpoint is the last non-missing measure from Week 12 to Week 34. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 0.35 (2.09)
Statistical Analysis 1: Comparison: Maintenance Arm; Null hypothesis is that duloxetine treatment effect on pain reduction in diabetic peripheral neuropathic pain (DPNP) is not maintained, as indicated by an increase of more than 1.5 point on the BPI 24-hour average pain scale. Null hypothesis is rejected at significance level 0.025 if the upper bound of one-sided 97.5% CI is less than or equal to non-inferiority margin of 1.5 point; Test type: Non-Inferiority or Equivalence — Non-inferiority margin of 1.5 point on the BPI 24-hour average pain scale; p < 0.001, t-test, 1 sided — Significance level 0.025; Mean Difference (Net) = 0.35, 97.5% CI [0.35 to 0.79]

2. Secondary Outcome: Maintenance Arm: Number of Patients With a ≥50% Reduction From Baseline (Week 0) in Brief Pain Inventory 24-hour Average Pain Item
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 0), Week 34
Population: Number of responders with a baseline and at least one non-missing post-baseline score. Endpoint is the last non-missing measure from Week 12 to Week 34. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
participants | 76

3. Secondary Outcome: Rescue Arm: Number of Patients With a ≥50% Reduction From Baseline (Week 0) in Brief Pain Inventory 24-hour Average Pain Item
Description: as for outcome 2
Time Frame: Baseline (Week 0), Week 34
Population: Number of non-responders with a baseline and at least one non-missing post-baseline score. Endpoint is the last non-missing measure from Week 12 to Week 34. Last observation carried forward.
Measure: Number; unit: participants
Arm/Group | Rescue Arm
Number analyzed (Participants) | 66
participants | 21

4. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Worst Pain Score at Week 34 Endpoint
Description: A self-reported scale that measures the severity of pain based on the worst pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 0.29 (2.78)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.269, t-test, 2 sided

5. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Worst Pain Score at Week 34 Endpoint
Description: as for outcome 4
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 67
units on a scale | -1.33 (2.96)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Least Pain Score at Week 34 Endpoint
Description: A self-reported scale that measures the severity of pain based on the least pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 0.24 (1.79)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.160, t-test, 2 sided

7. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Least Pain Score at Week 34 Endpoint
Description: as for outcome 6
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 67
units on a scale | -0.93 (3.07)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

8. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Average Pain Score at Week 34 Endpoint
Description: A self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 0.35 (2.09)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.075, t-test, 2 sided

9. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Average Pain Score at 34 Week Endpoint
Description: as for outcome 8
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 66
units on a scale | -1.39 (2.57)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Pain Right Now Score at Week 34 Endpoint
Description: A self-reported scale that measures the severity of pain based on the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 0.48 (2.28)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.026, t-test, 2 sided

11. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Pain Right Now Score at Week 34 Endpoint
Description: as for outcome 10
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 67
units on a scale | -1.12 (3.49)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.011, t-test, 2 sided

12. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: General Activity at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on general activity. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.22 (2.73)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.406, t-test, 2 sided

13. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: General Activity at Week 34 Endpoint
Description: as for outcome 12
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -1.01 (3.53)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.021, t-test, 2 sided

14. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Mood at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on mood. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.39 (2.63)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.124, t-test, 2 sided

15. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Mood at Week 34 Endpoint
Description: as for outcome 14
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -0.29 (3.62)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.505, t-test, 2 sided

16. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Walking Ability at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on walking ability. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.59 (3.22)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.058, t-test, 2 sided

17. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Walking Ability at 34 Week Endpoint
Description: as for outcome 16
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -1.15 (3.49)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.009, t-test, 2 sided

18. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Normal Work at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on normal work. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.63 (2.72)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

19. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Normal Work at Week 34 Endpoint
Description: as for outcome 18
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 67
units on a scale | -0.97 (3.40)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.022, t-test, 2 sided

20. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Relations With Other People at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on relations with other people. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.13 (2.22)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.550, t-test, 2 sided

21. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Relations With Other People at Week 34 Endpoint
Description: as for outcome 20
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 67
units on a scale | -0.12 (3.08)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.752, t-test, 2 sided

22. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Sleep at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on sleep. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | -0.10 (2.83)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.713, t-test, 2 sided

23. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Sleep at Week 34 Endpoint
Description: as for outcome 22
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -0.84 (3.69)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.066, t-test, 2 sided

24. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Enjoyment of Life at Week 34 Endpoint
Description: A self-reported scale that measures the interference of pain in the past 24 hours on enjoyment of life. The Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.11 (3.06)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.711, t-test, 2 sided

25. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Interference Score: Enjoyment of Life at Week 34 Endpoint
Description: as for outcome 24
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | 0.19 (3.79)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.678, t-test, 2 sided

26. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Brief Pain Inventory Average Interference at Week 34 Endpoint
Description: A self-reported scale that measures interference of pain on average of the 7 questions assessing the interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 111
units on a scale | 0.28 (2.34)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.216, t-test, 2 sided

27. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Brief Pain Inventory Average Interference at Week 34 Endpoint
Description: as for outcome 26
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -0.59 (3.04)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.113, t-test, 2 sided

28. Secondary Outcome: Maintenance Arm: Patient's Global Impressions of Improvement (PGI-I) at Week 34 Endpoint
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: Week 34
Population: Number of responders with at least one non-missing post-baseline score. Endpoint is the last non-missing measure from Week 12 to Week 34. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | 2.32 (1.33)

29. Secondary Outcome: Rescue Arm: Patient's Global Impressions of Improvement (PGI-I) at Week 34 Endpoint
Description: as for outcome 28
Time Frame: Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | 3.04 (1.32)

30. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Clinical Global Impressions of Severity (CGI-S) at Week 34 Endpoint
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 114
units on a scale | -0.11 (1.24)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.368, t-test, 2 sided

31. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Clinical Global Impressions of Severity (CGI-S) at Week 34 Endpoint
Description: as for outcome 30
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -0.46 (1.23)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.003, t-test, 2 sided

32. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Sensory Portion of the Short-Form McGill Pain Questionnaire at Week 34 Endpoint
Description: This instrument consists of 11 pain descriptors. The sensory pain portion scores range from 0 (none) to 3 (severe).
Time Frame: Baseline (Week 8), Week 34
Population: Number of responders with a baseline and ate least one non-missing post-baseline score. Endpoint is the last non-missing measure from Week 12 to Week 34. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 108
units on a scale | 0.31 (7.34)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.666, t-test, 2 sided

33. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Sensory Portion of the Short-Form McGill Pain Questionnaire at Week 34 Endpoint
Description: This instrument consists of 11 pain descriptors. The sensory pain portion scores range from 0 (none) to 3 (severe).
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -1.38 (7.60)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.138, t-test, 2 sided

34. Secondary Outcome: Maintenance Arm: Change From Baseline (Week 8) in Beck Depression Inventory-II (BDI-II) Total Score at Week 34 Endpoint
Description: A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maintenance Arm
Number analyzed (Participants) | 109
units on a scale | -0.82 (5.80)
Statistical Analysis 1: Comparison: Maintenance Arm; Test type: Superiority or Other; p = 0.145, t-test, 2 sided

35. Secondary Outcome: Rescue Arm: Change From Baseline (Week 8) in Beck Depression Inventory-II (BDI-II) Total Score at Week 34 Endpoint
Description: as for outcome 34
Time Frame: Baseline (Week 8), Week 34
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rescue Arm
Number analyzed (Participants) | 68
units on a scale | -0.53 (6.62)
Statistical Analysis 1: Comparison: Rescue Arm; Test type: Superiority or Other; p = 0.512, t-test, 2 sided

36. Secondary Outcome: Number of Participants Discontinuing in the Acute Phase
Time Frame: Baseline (Week 0) to Week 8
Population: Participants in Acute Phase (through Week 8).
Measure: Number; unit: participants
Arm/Group | Acute Phase
Number analyzed (Participants) | 216
participants
  Initiating at Week 0 | 216
  Continuing at Week 1 | 201
  Continuing at Week 8 | 184

37. Secondary Outcome: Number of Participants Discontinuing in Maintenance / Rescue Phase
Time Frame: Baseline (Week 8) to Week 34
Population: Participants in Maintenance / Rescue Phase (beyond Week 8 through Week 34)
Measure: Number; unit: participants
Groups:
- All Maintenance / Rescue Participants: Total of the Maintenance (No Dose Increase), Maintenance (Later Dose Increase) and Rescue arms. Depending on the group the patient was in, they either received duloxetine 60 mg once daily; 60 mg once daily and then increased to 120 mg once daily; or 120 mg once daily.
- Maintenance Arm (No Dose Increase): duloxetine 60 mg once daily
- Maintenance Arm (Later Dose Increase): duloxetine 60 mg once daily and then increasing to 120 mg once daily
- Rescue Arm: duloxetine 120 mg once daily
Arm/Group | All Maintenance / Rescue Participants | Maintenance Arm (No Dose Increase) | Maintenance Arm (Later Dose Increase) | Rescue Arm
Number analyzed (Participants) | 184 | 103 | 12 | 69
participants
  Entering at Week 8 | 184 | 103 | 12 | 69
  Continuing at Week 12 | 171 | 96 | 12 | 63
  Continuing at Week 16 | 142 | 92 | 11 | 39
  Continuing at Week 24 | 128 | 84 | 10 | 34
  Completing at Week 34 | 119 | 77 | 9 | 33

38. Secondary Outcome: Change From Baseline in Vital Signs: Heart Rate at Week 34 Endpoint
Time Frame: Baseline (Week 0), Week 34
Population: All patients who received either 60 mg or 120 mg duloxetine once daily.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Duloxetine 60 mg: Duloxetine: 60 milligrams once daily
- Duloxetine 120 mg: Duloxetine: 120 milligrams once daily
Arm/Group | Duloxetine 60 mg | Duloxetine 120 mg
Number analyzed (Participants) | 214 | 80
beats per minute | 2.4 (10.78) | 0.4 (11.46)

39. Secondary Outcome: Change From Baseline (Week 0) in Vital Signs: Diastolic Blood Pressure at Week 34 Endpoint
Time Frame: Baseline (Week 0), Week 34
Population: All patients who received either 60 mg or 120 mg duloxetine once daily.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine 60 mg | Duloxetine 120 mg
Number analyzed (Participants) | 214 | 80
mm Hg | -0.1 (9.39) | -1.0 (9.18)

40. Secondary Outcome: Change From Baseline (Week 0) in Vital Signs: Systolic Blood Pressure at Week 34 Endpoint
Time Frame: Baseline (Week 0), Week 34
Population: All patients who received either 60 mg or 120 mg duloxetine once daily.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Duloxetine 60 mg | Duloxetine 120 mg
Number analyzed (Participants) | 214 | 80
mm Hg | -4.2 (14.94) | 0.7 (15.27)

41. Secondary Outcome: Change From Baseline (Week 0) in Vital Signs: Weight at Week 34 Endpoint
Time Frame: Baseline (Week 0), Week 34
Population: All patients who received either 60 mg or 120 mg duloxetine once daily.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Duloxetine 60 mg | Duloxetine 120 mg
Number analyzed (Participants) | 214 | 80
kilograms (kg) | -1.3 (4.17) | 0.2 (3.16)

ADVERSE EVENTS:
Time Frame: 34 Weeks
Description: There were 12 patients who began the maintenance dose group who had their dose increased to rescue dose of 120 mg QD at some point during the maintenance period. Adverse events reported were attributed to the dose the participant was on at the time of the event, therefore, the 12 participants were also included in the 120 mg QD group.
Arm/Group | Duloxetine 60 mg | Duloxetine 120 mg
Serious Adverse Events (participants affected / at risk) | 18/216 | 2/81
Other Adverse Events (participants affected / at risk) | 135/216 | 40/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60 mg (N=216) | Duloxetine 120 mg (N=81)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Viral labyrinthitis (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 60 mg (N=216) | Duloxetine 120 mg (N=81)
Vertigo (Ear and labyrinth disorders) | 9 (9) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 9 (9) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 13 (13) | 1 (1)
Nausea (Gastrointestinal disorders) | 41 (46) | 3 (3)
Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2)
Asthenia (General disorders) | 11 (12) | 1 (1)
Chills (General disorders) | 7 (8) | 0 (0)
Fatigue (General disorders) | 11 (18) | 0 (0)
Influenza (Infections and infestations) | 5 (5) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 12 (12) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (9) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (15) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 2 (2)
Dizziness (Nervous system disorders) | 7 (9) | 1 (1)
Headache (Nervous system disorders) | 11 (24) | 3 (3)
Somnolence (Nervous system disorders) | 18 (19) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 1 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 7 (7) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 (16) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days